CLINICAL TRIAL: NCT06454929
Title: Comparison Between Operative And Non-operative Treatment of Displaced Medial Epicondyle Fractures In Children
Brief Title: Treatment of Displaced Medial Epicondyle Fractures In Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed ezzat mohamed eltaweel, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Medial Epicondyle Fracture
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Fractures, Bone
Keywords: medial epicondyle fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: operative by k-wires or screws or non-operative by cast immobilisation treatment (using randomization tables/software
Who Masked: Outcomes Assessor
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- operative group (Active Comparator): fixation by k-wires or screws
  Interventions: Procedure: operative
- non operative group (Active Comparator): fixation by cast immobilisation
  Interventions: Procedure: non-operative

INTERVENTIONS:
Procedure: operative — open reduction : fixation by k-wires or screws
  Arms: operative group
Procedure: non-operative — close reduction : by cast Immobilization
  Arms: non operative group

SUMMARY:
Compare the outcome of the operative and non-operative treatment; for fractures of the medial epicondyle of humerus in children as regards union, alignment and complications.

DETAILED DESCRIPTION:
On the distal humerus, posteromedially, is where the medial epicondyle apophysis is situated. It serves as the starting point for the flexor-pronator muscle and the ulnar collateral ligament. 12-20% of pediatric elbow fractures have been reported to be caused by fractures of the medial humeral epicondyle. Thirty to fifty percent of these fractures result in elbow dislocation, and eighteen to twenty percent of the fracture fragments become lodged in the elbow joint. The medial epicondyle fractures typically happen between the ages of 9 and 14 due to the insufficient ossification of the bone, which makes it more prone to failure early than the stronger soft-tissue attachments.

Optimal treatment for pediatric medial epicondyle fractures continues to be a topic of debate.

In the face of technical advancements, evolving surgical indications, and societal pressures, there is little concrete data demonstrating the superiority of either operative or non-operative treatment.

When a child's medial humeral epicondyle fracture is minimally displaced (less than 2 mm), non-operative therapy is recommended. The PedsQL Pediatric discomfort Questionnaire revealed that children who received non-operative treatment experienced reduced discomfort (3 vs. 15, p = 0.01) and had superior cosmetic results. There is a great deal of disagreement about how to treat displaced fractures (3-15 mm), with some surgeons supporting internal fixation as the non-union rate drops significantly. For upper-extremity athletes who need elbow stability to play their sport, surgery is also advised. Furthermore, it has been proposed that there are no statistically significant variations in outcomes between surgical and non-operative groups.

Fractures of the medial humeral epicondyle in children heal well with 3-4 weeks' immobilization. There is no common consensus in treatment of closed medial epicondyle fractures with >2 mm displacement (without incarceration of the fragment inside the joint or ulnar nerve dysfunction) that Open reduction and screw fixation improve outcome.

The purpose of our study is to compare the treatment outcomes and complications between operatively and non-operatively treated displaced medial epicondyle fractures. We aim to improve our understanding of the outcomes of these fractures to make treatment recommendations. We hypothesise that there is no difference in treatment outcomes between non-operative and operative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients Age < 16 years presenting with a ≥2 mm displaced non-incarcerated medial epicondyle fracture with or without concomitant elbow dislocation and normal ulnar nerve function.
* Acute fractures were defined as less than7 days between the date of injury and initiation of treatment

Exclusion Criteria:

* systemic bone disease
* concomitant fracture or injury of the same upper limb requiring operative intervention
* Open fractures, incarceration of the fragment inside the joint or ulnar nerve dysfunction require surgery

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The disabilities of the arm, shoulder and hand (QuickDASH) score | baseline
  QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.

REFERENCES:
- [Background] Pathy R, Dodwell ER. Medial epicondyle fractures in children. Curr Opin Pediatr. 2015 Feb;27(1):58-66. doi: 10.1097/MOP.0000000000000181. PMID 25564187
- [Background] Beck JJ, Bowen RE, Silva M. What's New in Pediatric Medial Epicondyle Fractures? J Pediatr Orthop. 2018 Apr;38(4):e202-e206. doi: 10.1097/BPO.0000000000000902. PMID 27861213
- [Background] Axibal DP, Carry P, Skelton A, Mayer SW. No Difference in Return to Sport and Other Outcomes Between Operative and Nonoperative Treatment of Medial Epicondyle Fractures in Pediatric Upper-Extremity Athletes. Clin J Sport Med. 2020 Nov;30(6):e214-e218. doi: 10.1097/JSM.0000000000000666. PMID 30277893